CLINICAL TRIAL: NCT03713710
Title: Self-Sampling for HPV Testing in African American Women - Mississippi Delta
Brief Title: Self-Sampling for Human Papillomavirus (HPV) Testing in African American Women - Mississippi Delta
Acronym: HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Isabel Scarinci, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: X161101004
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Cervical Cancer
Keywords: self-sampling for HPV testing
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Vaginal Smears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pap testing (Experimental): Women assigned to this arm will be scheduled a Pap testing appointment at the local health department
  Interventions: Behavioral: Pap testing
- Choice (Experimental): Women assigned to this arm will be given a choice between scheduling an appointment for a Pap testing at the health department or engage in self-sampling for HPV testing at home
  Interventions: Behavioral: Choice

INTERVENTIONS:
Behavioral: Pap testing — Women will be approached in the community by a Peer Health Educator and scheduled an appointment for a Pap testing at the local health department
  Arms: Pap testing
Behavioral: Choice — Women will be approached in the community by a Peer Health Educator and they will be given a choice between scheduling an appointment for a Pap testing at the local health department or engage in self-sampling for HPV testing at home
  Arms: Choice

SUMMARY:
The purpose of this study is to examine the efficacy and costs of this patient-centered approach ("Choice" between two cervical cancer screening modalities) in adherence to cervical cancer screening as compared to the current standard of care within the public health system in Mississippi (Pap test at the local department -"Pap") among un/under-screened African American women in the Mississippi Delta using a theory-based, culturally relevant intervention implemented by Peer Health Educators (PHEs).

DETAILED DESCRIPTION:
OBJECTIVE: Our objective is to examine the efficacy and costs of a patient-centered approach ("Choice" between self-sampling and Pap test) in adherence to cervical cancer screening as compared to Pap test at the local health department ("Pap") among un/under-screened African American women in the Mississippi Delta.

HYPOTHESES: Women in the "Choice" arm will have a higher cervical cancer screening adherence as well as higher satisfaction than women assigned to the "Pap" arm; (2) Within the "Choice" arm, more women will choose and complete self-sampling than Pap test; and (3) The "Choice" intervention will be on average less costly and more cost-effective than the "Pap" intervention.

SPECIFIC AIMS: (1) To compare the impact of these two intervention approaches, "Choice" versus "Pap", on cervical cancer screening adherence through a group randomized controlled trial; (2) To compare patient satisfaction between the two intervention approaches; and (3) To compare the costs and cost-effectiveness of these two intervention approaches, "Choice" versus "Pap".

STUDY DESIGN: 12 towns will be randomized to either "Choice" or "Pap" (180 women/arm). Peer Health Educators (PHEs) will identify African American women who report not having undergone cervical cancer screening in the past three years and deliver a brief theory-based, cultural relevant educational session on cervical cancer and screening using a door-to-door approach. Women randomized to the "Pap" arm will be provided with information on how to schedule an appointment at the local health department. Women randomized to the "Choice" arm will be given the choice of attending the health department for a Pap test or self-collecting their own sample at home to be sent for HPV testing. PHEs will follow-up with women in either arm who have a positive test in order to assure diagnostic evaluation and care.

ELIGIBILITY:
Inclusion Criteria:

* no personal history of cervical cancer
* not have engaged in cervical cancer screening in the past four years

Exclusion Criteria:

* none

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 335 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
adherence to cervical cancer screening | baseline to 30 days
  adherence to cerivcal cancer screening by attending the Pap testing or returning the self-collected sample for HPV testing

SECONDARY OUTCOMES:
Satisfaction with the intervention | baseline to 6 months
  We will assess participants' satisfaction with intervention through self-report (satisfaction questionnaire - satisfied/very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel C. Scarinci, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Mississippi State Department of Health, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scarinci IC, Li Y, Tucker L, Campos NG, Kim JJ, Peral S, Castle PE. Given a choice between self-sampling at home for HPV testing and standard of care screening at the clinic, what do African American women choose? Findings from a group randomized controlled trial. Prev Med. 2021 Jan;142:106358. doi: 10.1016/j.ypmed.2020.106358. Epub 2020 Dec 16. PMID 33338505